CLINICAL TRIAL: NCT02021500
Title: MPACT Extension Study: Multicenter, Survival Data Collection in Subjects Previously Enrolled in Protocol CA046
Brief Title: A Study to Collect Survival Data on Patients Previously Enrolled in Abraxane Pancreatic Cancer Study CA046.
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: ABI-007-PANC-CA046C
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients previously enrolled in study CA046: No intervention is being given in this extension study which is gathering survival information on participants of study NCT 00844649 (Celgene study CA046) who were known to be alive as of March 2013)
  Interventions: Drug: ABI-007

INTERVENTIONS:
Drug: ABI-007 — No intervention is being given in this extension study which is gathering survival information on participants of study NCT 00844649 (Celgene study CA046) who were known to be alive as of March 2013)

SUMMARY:
A study to collect survival data on patients previously enrolled in Abraxane pancreatic cancer study CA046.

DETAILED DESCRIPTION:
A study to collect survival status of CA046 subjects who were know to be alive at the last report of vital status for CA046 - approximate timeframe - end of March, 2013. Once consent is given, on a quarterly basis, information on status will be collected to include:

* Vital Status
* Date of disease progression
* Subsequent anticancer therapy for pancreatic adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Must have been enrolled in the CA046 study Must have been living at the time of the last survival follow-up (approximate timeframe - end of March, 2013) Must understand and be able to give informed consent (if a subject is deceased, proper legal consent (ie, next of kin, legal representative) will be obtained prior to collection of data)

Exclusion Criteria:

* Consent refused for any reason

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients previously enrolled in study CA046
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-01-02 (Actual); Primary Completion 2015-04-16 (Actual); Study Completion 2015-04-16 (Actual)

PRIMARY OUTCOMES:
Overall Survival | up to 3 years
  Number of participants who survive

SECONDARY OUTCOMES:
Disease progression | up to 3 years
  Date of disease progression and subsequent anticancer therapy for pancreatic adenocarcinoma other than that already recorded for subject while enrolled in CA046

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Manax, MD, Study Director — Celgene
Locations (39):
- United States (16):
  - TGen Clinical Research Services, Scottsdale, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Pacific Shores Medical Group, Long Beach, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Florida Cancer Specialists, Englewood, Florida
  - Florida Cancer Specialist, Tavares, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Arena Oncology Associates, Lake Success, New York
  - UPMC Cancer Pavillion, Pittsburgh, Pennsylvania
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - South Texas Oncology and Hematology (STOH), San Antonio, Texas
  - Fairfax-Northern Virginia Haematology-Oncology, Fairfax, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Froedtert and Medical College ID Clinic, Milwaukee, Wisconsin
- Australia (4):
  - Macarthur Cancer Therapy Centre, Campbelltown, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - HOCA - the Wesley Clinic for Heamatology and Oncology, Auchenflower, Queensland
  - Mater Medical Center, South Brisbane
- Austria (3):
  - Landesklinikum St. Pölten, Sankt Pölten
  - Medizinische Universität Wien, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Centre Hospsitalier Universitaire de Montreal - Notre Dame, Montreal, Quebec
- France (2):
  - Hôpital Beaujon, Clichy
  - Hôpital Saint Antoine, Paris
- Germany (2):
  - Kliniken Essen-Mitte, Essen
  - LMU Klinikum der Universität München, München
- Italy (4):
  - Ospedale San Raffaele S.r.l., Milan
  - Azienda Ospedaliera Niguarda Cà Granda, Milan
  - Ospedale Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotundo
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Municipal institution Multifield City Clinical Hospital #4 of Dnipropetrovsk Regional Council, Dnipropetrovsk, Ukraine

REFERENCES:
- [Background] Ramanathan RK, Goldstein D, Korn RL, Arena F, Moore M, Siena S, Teixeira L, Tabernero J, Van Laethem JL, Liu H, McGovern D, Lu B, Von Hoff DD. Positron emission tomography response evaluation from a randomized phase III trial of weekly nab-paclitaxel plus gemcitabine versus gemcitabine alone for patients with metastatic adenocarcinoma of the pancreas. Ann Oncol. 2016 Apr;27(4):648-53. doi: 10.1093/annonc/mdw020. Epub 2016 Jan 22. PMID 26802153
- [Background] Chiorean EG, Von Hoff DD, Reni M, Arena FP, Infante JR, Bathini VG, Wood TE, Mainwaring PN, Muldoon RT, Clingan PR, Kunzmann V, Ramanathan RK, Tabernero J, Goldstein D, McGovern D, Lu B, Ko A. CA19-9 decrease at 8 weeks as a predictor of overall survival in a randomized phase III trial (MPACT) of weekly nab-paclitaxel plus gemcitabine versus gemcitabine alone in patients with metastatic pancreatic cancer. Ann Oncol. 2016 Apr;27(4):654-60. doi: 10.1093/annonc/mdw006. Epub 2016 Jan 22. PMID 26802160
- [Background] Goldstein D, Von Hoff DD, Moore M, Greeno E, Tortora G, Ramanathan RK, Macarulla T, Liu H, Pilot R, Ferrara S, Lu B. Development of peripheral neuropathy and its association with survival during treatment with nab-paclitaxel plus gemcitabine for patients with metastatic adenocarcinoma of the pancreas: A subset analysis from a randomised phase III trial (MPACT). Eur J Cancer. 2016 Jan;52:85-91. doi: 10.1016/j.ejca.2015.10.017. Epub 2015 Dec 1. PMID 26655559
- [Background] Portal A, Pernot S, Tougeron D, Arbaud C, Bidault AT, de la Fouchardiere C, Hammel P, Lecomte T, Dreanic J, Coriat R, Bachet JB, Dubreuil O, Marthey L, Dahan L, Tchoundjeu B, Locher C, Lepere C, Bonnetain F, Taieb J. Nab-paclitaxel plus gemcitabine for metastatic pancreatic adenocarcinoma after Folfirinox failure: an AGEO prospective multicentre cohort. Br J Cancer. 2015 Sep 29;113(7):989-95. doi: 10.1038/bjc.2015.328. Epub 2015 Sep 15. PMID 26372701
- [Background] Goldstein D, El-Maraghi RH, Hammel P, Heinemann V, Kunzmann V, Sastre J, Scheithauer W, Siena S, Tabernero J, Teixeira L, Tortora G, Van Laethem JL, Young R, Penenberg DN, Lu B, Romano A, Von Hoff DD. nab-Paclitaxel plus gemcitabine for metastatic pancreatic cancer: long-term survival from a phase III trial. J Natl Cancer Inst. 2015 Jan 31;107(2):dju413. doi: 10.1093/jnci/dju413. Print 2015 Feb. PMID 25638248
- [Background] Vogel A, Pelzer U, Salah-Eddin AB, Koster W. First-line nab-paclitaxel and gemcitabine in patients with metastatic pancreatic cancer from routine clinical practice. In Vivo. 2014 Nov-Dec;28(6):1135-40. PMID 25398812
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Al-Hajeili M, Azmi AS, Choi M. Nab-paclitaxel: potential for the treatment of advanced pancreatic cancer. Onco Targets Ther. 2014 Feb 4;7:187-92. doi: 10.2147/OTT.S40705. eCollection 2014. PMID 24523592
- [Background] Tabernero J, Chiorean EG, Infante JR, Hingorani SR, Ganju V, Weekes C, Scheithauer W, Ramanathan RK, Goldstein D, Penenberg DN, Romano A, Ferrara S, Von Hoff DD. Prognostic factors of survival in a randomized phase III trial (MPACT) of weekly nab-paclitaxel plus gemcitabine versus gemcitabine alone in patients with metastatic pancreatic cancer. Oncologist. 2015 Feb;20(2):143-50. doi: 10.1634/theoncologist.2014-0394. Epub 2015 Jan 12. PMID 25582141
- [Background] Chiorean EG, Von Hoff DD, Tabernero J, El-Maraghi R, Ma WW, Reni M, Harris M, Whorf R, Liu H, Li JS, Manax V, Romano A, Lu B, Goldstein D. Second-line therapy after nab-paclitaxel plus gemcitabine or after gemcitabine for patients with metastatic pancreatic cancer. Br J Cancer. 2016 Jul 12;115(2):188-94. doi: 10.1038/bjc.2016.185. Epub 2016 Jun 28. PMID 27351217
- [Background] Tehfe M, Dowden S, Kennecke H, El-Maraghi R, Lesperance B, Couture F, Letourneau R, Liu H, Romano A. nab-Paclitaxel Plus Gemcitabine Versus Gemcitabine in Patients with Metastatic Pancreatic Adenocarcinoma: Canadian Subgroup Analysis of the Phase 3 MPACT Trial. Adv Ther. 2016 May;33(5):747-59. doi: 10.1007/s12325-016-0327-4. Epub 2016 Apr 16. PMID 27085323
- [Background] Scheithauer W, Ramanathan RK, Moore M, Macarulla T, Goldstein D, Hammel P, Kunzmann V, Liu H, McGovern D, Romano A, Von Hoff DD. Dose modification and efficacy of nab-paclitaxel plus gemcitabine vs. gemcitabine for patients with metastatic pancreatic cancer: phase III MPACT trial. J Gastrointest Oncol. 2016 Jun;7(3):469-78. doi: 10.21037/jgo.2016.01.03. PMID 27284481
- [Background] Vogel A, Rommler-Zehrer J, Li JS, McGovern D, Romano A, Stahl M. Efficacy and safety profile of nab-paclitaxel plus gemcitabine in patients with metastatic pancreatic cancer treated to disease progression: a subanalysis from a phase 3 trial (MPACT). BMC Cancer. 2016 Oct 21;16(1):817. doi: 10.1186/s12885-016-2798-8. PMID 27769210
- [Background] Tabernero J, Kunzmann V, Scheithauer W, Reni M, Shiansong Li J, Ferrara S, Djazouli K. nab-Paclitaxel plus gemcitabine for metastatic pancreatic cancer: a subgroup analysis of the Western European cohort of the MPACT trial. Onco Targets Ther. 2017 Feb 2;10:591-596. doi: 10.2147/OTT.S124097. eCollection 2017. PMID 28203092
- [Background] Kunzmann V, Ramanathan RK, Goldstein D, Liu H, Ferrara S, Lu B, Renschler MF, Von Hoff DD. Tumor Reduction in Primary and Metastatic Pancreatic Cancer Lesions With nab-Paclitaxel and Gemcitabine: An Exploratory Analysis From a Phase 3 Study. Pancreas. 2017 Feb;46(2):203-208. doi: 10.1097/MPA.0000000000000742. PMID 27841795